CLINICAL TRIAL: NCT05855967
Title: A 24-Week Multicenter, Open-label, Single-arm, Phase 4 Study to Evaluate the Safety of Ixekizumab in Patients With Moderate-to-Severe Plaque Psoriasis or Active Psoriatic Arthritis in India
Brief Title: A Study of Ixekizumab (LY2439821) in Participants Aged ≥18 Years With Moderate-to-Severe Plaque or Active Psoriatic Arthritis in India
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18528; I1F-IN-RHCZ (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Plaque Psoriasis; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — ixekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ixekizumab - PsO With no Active PsA (Experimental): Participants with plaque psoriasis (PsO) with no active psoriatic arthritis (PsA) received:
  * Ixekizumab 160 milligram (mg) subcutaneous (SC) injection as loading dose at Week 0, followed by;
  * Ixekizumab 80 mg SC injection every 2 weeks (Q2W) at Week 2, 4, 6, 8, and 10
  * Ixekizumab 80 mg SC injection every 4 weeks (Q4W) at Week 12, 16, and 20
  Interventions: Drug: Ixekizumab
- Ixekizumab - Active PsA (Experimental): Participants with active psoriatic arthritis (PsA) with moderate to severe plaque psoriasis (PsO) received:
  * Ixekizumab 160 mg SC injection as loading dose at Week 0, followed by;
  * Ixekizumab 80 mg SC injection Q2W at Week 2, 4, 6, 8, and 10
  * Ixekizumab 80 mg SC injection Q4W at Week 12, 16, and 20
  Participants with active PsA without moderate to severe PsO received:
  * Ixekizumab 160 mg SC injection as loading dose at Week 0, followed by
  * Ixekizumab 80 mg SC injection Q4W at Week 4, 8, 12, 16, and 20.
  Interventions: Drug: Ixekizumab

INTERVENTIONS:
Drug: Ixekizumab — Administered SC
  Other Names: LY2439821

SUMMARY:
The main purpose of this study is to investigate the safety and tolerability of ixekizumab in participants in India with moderate-to-severe plaque psoriasis (PsO) or active psoriatic arthritis (PsA)

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Male or nonpregnant, nonbreastfeeding female participants.

For PsO Participants:

* Present with chronic PsO based on a confirmed diagnosis of chronic PsO vulgaris for at least 6 months prior to baseline
* Have ≥10% Body Surface Area (BSA) of psoriasis at screening (Visit 1) and baseline
* Have both an static Physician's Global Assessment (sPGA) score of ≥3 and Psoriasis Area and Severity Index (PASI) score ≥12 at screening and baseline

For PsA Participants

* Have a diagnosis of active PsA for at least 6 months (based on a detailed medical history provided by the patient, and a physical exam by the Study Investigator, and/or other evidence such as that provided by joint x-rays, that establishes a history consistent with a diagnosis of active PsA of at least 6 months' duration) and currently meet the Classification for PsA (CASPAR) criteria.
* Have active PsA defined as the presence of at least 3/68 tender and at least 3/66 swollen joints, as determined by the Tender and Swollen Joint Count Assessment Form at screening and baseline.
* Presence of active PsO or a documented history of psoriasis.

Exclusion Criteria:

* Have previously completed or withdrawn from this study, participated in any other study with ixekizumab, or have participated in any study investigating other IL-17 antagonists.
* Have a history of drug-induced PsO.
* Have a known allergy or hypersensitivity to any biologic therapy that would pose an unacceptable risk to the patient if participating in this study.
* Had any major surgery within 8 weeks prior to baseline (Week 0; Visit 2), or will require such during the study that, in the opinion of the investigator in consultation with Lilly or its designee, would pose an unacceptable risk to the participant
* Have diagnosis or history of malignant disease within the 5 years prior to baseline
* Have any other active or recent infection within 4 weeks of baseline

For PsO Participants:

* Have received systemic non-biologic PsO therapy (within 4 weeks prior to baseline)
* Have pustular, erythrodermic, and/or guttate forms of PsO
* Had a clinically significant flare of PsO during the 12 weeks prior to baseline (Week 0).
* Have allergy to rubber or latex.

For PsA Participants:

* Have used conventional synthetic disease-modifying antirheumatic drug (csDMARDs) other than methotrexate (MTX), leflunomide, sulfasalazine, or cyclosporine in the 8 weeks prior to baseline
* Have received treatment with interleukin (IL)17 or IL-12/23 targeted Mab therapy
* Are currently receiving treatment with any biologic or small molecule therapy for PsA or PsO, including investigational therapies (such as, but not limited to, a tumor necrosis factor inhibitor (TNFi), IL-1 receptor antagonists, IL-6 inhibitor, anti-IL12/23p40, T cell or B cell targeted therapies, phosphodiesterase (PDE) 4 inhibitors, or Janus Kinase (JAK) inhibitors), or have received denosumab.
* Have had surgical treatment of a joint within 8 weeks prior to baseline or will require such up to Week 24.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- India (14):
  - King George Hospital, Vizag, Andhra Pradesh
  - All India Institute of Medical Sciences, Raipur, Chhattisgarh
  - V.S. General Hospital, Ahmedabad, Gujarat
  - Amber Clinic, Ahmedabad, Gujarat
  - B. J. Medical College & Civil Hospital, Ahmedabad, Gujarat
  - GMERS Medical College & Hospital, Ahmedabad, Gujarat
  - Tristar Hospital, Surat, Gujarat
  - Father Muller Medical College Hospital, Mangalore, Karnataka
  - Dr. D. Y. Patil Medical College & Hospital, Navi Mumbai, Maharashtra
  - Grant Medical Foundation - Ruby Hall Clinic, Pune, Maharashtra
  - Oyster & Pearl Hospitals (Phadnis Clinic Pvt. Ltd.), Pune, Maharashtra
  - Postgraduate Institute of Medical Education & Research, Chandigarh, Punjab
  - Wizderm Specialty Skin And Hair Clinic, Kolkata, West Bengal
  - Medical College & Hospital, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ixekizumab - PsO With no Active PsA | Ixekizumab - Active PsA
Started | 150 | 100 (* PsA participants with PsO = 59 * PsA participants without PsO = 41)
Received at Least One Dose of Study Drug | 150 | 100
Q2W/Q4W Ixekizumab Dosing Regimen | 150 | 59
Q4W Ixekizumab Dosing Regimen | 0 | 41
Completed | 141 | 94
Not Completed | 9 | 6
Not completed — Withdrawal by Subject | 7 | 5
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study treatment.
Groups:
- Ixekizumab - PsO With no Active PsA: Participants with plaque psoriasis (PsO) with no active psoriatic arthritis (PsA) received:
  * Ixekizumab 160 mg SC injection as loading dose at Week 0, followed by;
  * Ixekizumab 80 mg SC injection Q2W at Week 2, 4, 6, 8, and 10
  * Ixekizumab 80 mg SC injection Q4W at Week 12, 16, and 20
- Total: Total of all reporting groups
Arm/Group | Ixekizumab - PsO With no Active PsA | Ixekizumab - Active PsA | Total
Number analyzed (Participants) | 150 | 100 | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 141 | 92 | 233
  >=65 years | 9 | 8 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 33 | 61
  Male | 122 | 67 | 189
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 20 | 28
  Unknown or Not Reported | 142 | 80 | 222
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 150 | 100 | 250
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  India | 150 | 100 | 250

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs), and Treatment Emergent Adverse Events (TEAEs) and AEs of Special Interests (AESIs) From Week 0 to Week 24
Description: * An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria listed: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect.
  * TEAE is defined as an event that first occurred or worsened in severity after baseline and on or prior to the date of the last visit within the treatment period.
Time Frame: Week 0 to Week 24
Population: All participants who received at least 1 dose of study treatment. As per prespecified analysis in the statistical analysis plan, adverse events were collected and analyzed by ixekizumab dosing regimen [that is, Q2W/Q4W and Q4W].
Measure: Count of Participants; unit: Participants
Groups:
- Q2W/Q4W Ixekizumab Dosing Regimen: Participants from PsO With no Active PsA arm and Active PsA arm with moderate to severe plaque psoriasis (PsO) who received Q2W/Q4W Ixekizumab dosing regimen.
- Q4W Ixekizumab Dosing Regimen: Participants from Active PsA arm without moderate to severe PsO who received Q4W Ixekizumab dosing regimen.
Arm/Group | Q2W/Q4W Ixekizumab Dosing Regimen | Q4W Ixekizumab Dosing Regimen
Number analyzed (Participants) | 209 | 41
Participants
  SAEs | 1 | 0
  TEAEs | 60 | 8
  AESIs | 39 | 6

2. Secondary Outcome: PsO With no Active PsA: Percentage of Participants With PsO Achieving ≥75% Improvement From Baseline in Psoriasis Area and Severity Index (PASI-75) at Week 12
Description: Participants achieving a PASI-75 without the use of other background antipsoriasis therapy were considered responders. The PASI quantifies the severity of a psoriasis based on lesion severity and the percent of body surface area (BSA) affected. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The sum of severity scores for erythema, thickness, and scaling is multiplied by the degree of involvement for each anatomic region and then multiplied by a constant corresponding to the region's percent BSA (0.1, 0.3, 0.2, and 0.4 for the above 4 regions, respectively). The resultant score for each anatomic region is then summed to yield the final PASI score. It ranges from 0 to 72, with higher scores reflecting greater disease severity.
Time Frame: Week 12
Population: All participants with a psoriasis indication, who do not qualify for active psoriatic arthritis (PsA) and had received at least 1 dose of study treatment. As per planned analysis, the outcome measure was planned to be analyzed for participants with plaque psoriasis (PsO) and with no active psoriatic arthritis (PsA).
Measure: Number; unit: percentage of participant
Arm/Group | Ixekizumab - PsO With no Active PsA
Number analyzed (Participants) | 150
percentage of participant | 86.0

3. Secondary Outcome: PsO With no Active PsA: Percentage of PsO Participants With a Static Physician Global Assessment (sPGA) Score of 0 (Clear) or 1 (Minimal)
Description: The sPGA is an assessment by the physician to determine participant's overall psoriatic lesions, at a given time point. For the analysis of responses, the participant's psoriasis indication is assessed on a 5-point scale as: 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe) incorporating an assessment of the severity of the three primary signs of the disease: induration, erythema, and degree of scaling.
  The investigator examines all of the lesions on the participant and assigns a score ranging from 0 to 5 for induration, erythema and degree of scaling. Scores for induration, erythema and scaling are then summed, and the mean of these 3 scores produces the overall sPGA score.
  Participants with an sPGA score of 0 (clear) or 1 (minimal) were considered responders and are reported here.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Ixekizumab - PsO With no Active PsA
Number analyzed (Participants) | 150
percentage of participants | 65.3

4. Secondary Outcome: Active PsA: Percentage of Active Psoriatic Arthritis Participants Who Achieved 20% Improvement From Baseline in American College of Rheumatology 20 (ACR20) at Week 24
Description: The ACR 20 is defined as:
  * 20% improvement from baseline in both tender joint count (68 counts) and swollen joint count (66 counts)
  * 20% improvements improvement in at least three of the following five items: Patient's global assessment of arthritis pain (measured on a 100-mm visual analog scale [VAS]); Patient's global assessment of disease activity (measured on a 100-mm VAS); Physician's global assessment of disease activity (measured on a 100-mm VAS); Patient's assessment of physical function as measured by the Health Assessment Questionnaire - Disability Index (HAQ-DI); Acute-phase reactant as measured by high-sensitivity C-reactive protein (hs-CRP) assay.
Time Frame: Week 24
Population: All participants with an active psoriatic arthritis indication who received at least 1 dose of study treatment. As per planned analysis, the outcome measure was planned to be analyzed for participants with active psoriatic Arthritis.
Measure: Number; unit: percentage of participants
Arm/Group | Ixekizumab - Active PsA
Number analyzed (Participants) | 100
percentage of participants | 84.0

ADVERSE EVENTS:
Time Frame: Week 0 up to 36 Weeks
Description: All enrolled participants who received at least 1 dose of study treatment. As per prespecified analysis in the statistical analysis plan, adverse events were reported by Ixekizumab dosing regimen [that is, Q2W/Q4W and Q4W].
Groups:
- Q2W/Q4W Ixekizumab Dosing Regimen: Participants from PsO with no active PsA arm and active PsA arm with moderate to severe plaque psoriasis (PsO) received Q2W/Q4W Ixekizumab dosing regimen.
Arm/Group | Q2W/Q4W Ixekizumab Dosing Regimen | Q4W Ixekizumab Dosing Regimen
All-Cause Mortality (participants affected / at risk) | 0/209 | 0/41
Serious Adverse Events (participants affected / at risk) | 1/209 | 0/41
Other Adverse Events (participants affected / at risk) | 66/209 | 9/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Q2W/Q4W Ixekizumab Dosing Regimen (N=209) | Q4W Ixekizumab Dosing Regimen (N=41)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Q2W/Q4W Ixekizumab Dosing Regimen (N=209) | Q4W Ixekizumab Dosing Regimen (N=41)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 4 (4) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 18 (18) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Body tinea (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Latent tuberculosis (Infections and infestations) | 18 (18) | 4 (4)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Pyoderma (Infections and infestations) | 1 (1) | 0 (0)
Tinea cruris (Infections and infestations) | 3 (3) | 0 (0)
Typhoid fever (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT05855967/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT05855967/SAP_001.pdf